CLINICAL TRIAL: NCT02868138
Title: Evaluation of Clinical Effectiveness, Quality of Life, and Compliance in Patients With Sickle Cell Disease Receiving Hydroxyurea
Brief Title: Study of Hydroxyurea to Treat Sickle Cell Disease
Status: Completed | Type: Observational
Sponsor: Mersin University (Other)
Responsible Party: Principal Investigator, Bahar TUNCTAN, Prof. Dr., Mersin University
Other Study IDs: MEUKAEK-2016/27 - 16-AKD-19
Record Dates: First submitted 2016-08-08; First posted 2016-08-16 (Estimated); Last update posted 2016-08-16 (Estimated); Status verified 2016-08

CONDITIONS: Sickle Cell Disease
Keywords: Sickle cell disease; Hydroxyurea; Compliance
MeSH Terms: conditions — Anemia, Sickle Cell; Patient Compliance

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

SUMMARY:
The aim of this single-center observational study was to evaluate quality of life, clinical effectiveness, and satisfaction in pediatric and young adult patients with sickle cell disease receiving hydroxyurea.

DETAILED DESCRIPTION:
In this study, 34 pediatric (HbSS: n= 5; HbSβ0: n= 29) and 16 (HbSS: n=5; HbSβ0: n= 11) young adult adult patients with sickle cell disease receiving hydroxyurea for at least a year were participated. Upon receipt of Informed Consent Form, Case Report Form, Demographic Data Collection Form, Child Health Questionnaire-Parent Form, Life Quality Survey Short Form-36, and Hydroxyurea Therapy Satisfaction Survey were used to obtain data for effectiveness of hydroxyurea therapy and parameters that may affect compliance to treatment and life quality of the participants.

Regarding the normal ranges, ferritin, hemoglobin A, A2, F, and S, platelet, mean corpuscular volume, erythrocyte distribution width, basophil percentage, monocyte, monocyte percentage, total bilirubin, direct bilirubin, and C-reactive protein values were higher while hemoglobin, hematocrit, and erythrocyte values were lower in these patients. Our findings regarding quality of life and satisfaction with hydroxyurea therapy indicated that the patients with sickle cell disease had lower scores.

Demographic, clinical, and therapeutic variables as well as comorbid diseases and concomitant drug use when considered together, these findings suggest that the health quality and compliance of the pediatric and young adult patients to therapy might be low due to not sufficiently effective hydroxyurea therapy in addition to comorbidities, concomitant drug use, and side effects.

ELIGIBILITY:
Inclusion Criteria:

1. Patients willing to participate in the study
2. Pediatric and young adult patients
3. Patients diagnosed with HbSS or HbSβ0 sickle cell disease
4. Patients receiving hydroxyurea for at least a year.

Exclusion Criteria:

1. Patients not meeting the inclusion criteria
2. Patients not willing to participate in the study
3. Patients diagnosed with other types of anemia except HbSS or HbSβ0 sickle cell disease
4. Patients not receiving hydroxyurea for at least a year
5. Patients having other conditions such as physical and/or mental difficulties which may affect their quality of life
6. Patients having any contrindication against hydroxyurea

Ages: 7 Years to 22 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Study Population: Pediatric (7-17 years) and young adult (18-22 years) patients with sickle cell disease who received hydroxyurea
Sampling Method: Non-Probability Sample
Enrollment: 50 (Actual)
Dates: Start 2016-05; Primary Completion 2016-07 (Actual); Study Completion 2016-07 (Actual)

PRIMARY OUTCOMES:
Effectiveness and acceptance of hydroxyurea therapy in patients | Up to 12 weeks

SECONDARY OUTCOMES:
Demographic characteristics of patients using Demographic Data Collection Form | Up to 12 weeks
Clinical characteristics of patients using Case Report Form | Up to 12 weeks
Health status of pediatric patients using Child Health Questionnaire-Parent Form | Up to 12 weeks
Quality of life of young adult patients using Life Quality Survey Short Form-36 | Up to 12 weeks
Effectiveness of hydroxyurea therapy in patients using Case Report Form | Up to 12 weeks
Acceptance of hydroxyurea therapy in patients using Hydroxyurea Satisfaction Survey | Up to 12 weeks

CONTACTS AND LOCATIONS:
Overall Officials: BAHAR TUNCTAN, Ph.D., Study Chair — MERSIN UNIVERSITY FACULTY OF PHARMACY DEPARTMENT OF PHARMACOLOGY
Locations (1):
- Selma Unal, Mersin, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: Yes